CLINICAL TRIAL: NCT00981266
Title: Study of the Safety and Effectiveness of the Mentor Spectra/Becker 80 Adjustable Breast Implant in Subjects Who Are Undergoing Primary Augmentation or Augmentation Revision
Brief Title: Spectra Breast Implant Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision. Study never started
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A101-0501-10
Record Dates: First submitted 2009-07-28; First posted 2009-09-22 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Augmentation; Augmentation Revision; General Breast Enlargement; Post-lactational Involution; Asymmetry
Keywords: Augmentation; Augmentation Revision
MeSH Terms: interventions — Breast Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Augmentation (Other): The study population will consist of women aged 22 or over who are undergoing primary breast augmentation.
  The Augmentation cohort will include candidates for general breast enlargement, post-lactational involution and/or asymmetry.
  Interventions: Device: Mentor Spectra/Becker 80 Breast Implant
- Augmentation Revision (Other): The study population will consist of women aged 22 or over who are undergoing augmentation revision.
  The Augmentation Revision cohort will include candidates with previous augmentation with silicone-filled or saline-filled implants.
  Interventions: Device: Mentor Spectra/Becker 80 Breast Implant

INTERVENTIONS:
Device: Mentor Spectra/Becker 80 Breast Implant — The Mentor Smooth Spectra/Becker 80 Adjustable Breast Implant has a low bleed, gel-filled outer lumen and an adjustable saline-fillable inner lumen. The inner lumen can be gradually filled with saline over a period of time via the fill tube by injecting saline through the injection dome. Once filled to the desired volume, the fill tube and injection dome are removed, and the prosthesis remains in position as a breast implant. Its purpose is to provide volume flexibility and projection adjustability.
  Other Names: Breast Implant; Double Lumen Breast-Implant; Becker 80 Implant; Spectra Implant

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of Mentor's Spectra/Becker 80 Adjustable Breast Implants in women who are undergoing primary or revision breast augmentation. Safety information on the rate of complications, such as infection, will be collected and used to help determine device safety. These implants are investigational devices.

Approximately 450 patients at sites across the United States will be enrolled in this research study by up to 30 sites. These patients will be implanted with Spectra/Becker 80 implant and monitored for 10 years to collect information on risks associated with the implant surgery as well as changes in the way these patients feel about themselves.

DETAILED DESCRIPTION:
Silicone gel-filled breast implants were introduced in the early sixties and were in wide-scale distribution by the time the Medical Device Amendments to the Food Drug and Cosmetic Act was passed in 1976. In 1983, gel-filled breast implants were designated as Class III devices requiring premarket approval. In May 1990, the Food and Drug Administration (FDA) published a proposed request (515(b)) for Pre-market Approval Applications (PMA) and in April 1991 published the final request. This final publication put manufacturers of gel-filled breast implants on notice that for continued marketing of gel-filled breast implants, a PMA was due to FDA in 90 days from the final publication date.

A Pre-Market Approval (PMA) for the Mentor gel-filled breast implants was filed with the FDA in July 1991. At the FDA General and Plastic Surgery Advisory Committee meeting in November 1991, the committee recommended the submission of additional information to establish the safety and effectiveness of gel-filled breast implants.

In January 1992, the FDA Commissioner announced a voluntary moratorium of the sale of gel-filled breast implants to allow the advisory panel time to assess additional information. In April 1992, the moratorium was lifted but only for reconstruction and revision subjects. Every subject implanted had to be part of an Adjunct Study, in addition to being offered participation in a registry of gel-filled breast implant subjects. The Adjunct Study devices included the round MemoryGel, Becker Expander/Prosthesis and the Lumera implants. In order to be implanted with gel-filled implants for augmentation, women had to be enrolled in an Investigational Device Exemption (IDE) clinical trial.

A PMA for Mentor's MemoryGel™ Silicone Gel-Filled breast implants (which did not include the Becker Expander/Breast Implants) was subsequently filed with FDA in December 2003, and approved in November 2006 (P030053). As a condition of approval of P030053, new enrollment in Mentor's Adjunct Study has ceased, and women no longer have access to the Becker Expander/Breast Implants or any Adjustable Gel-Filled implants. The Spectra/Becker 80 Adjustable Breast Implants were not included in the Adjunct Study.

This study is designed to study the safety and effectiveness of Mentor's Spectra/Becker 80 Adjustable Breast Implants for primary breast augmentation or augmentation revision.

ELIGIBILITY:
Inclusion Criteria:

* Subject is genetic female and is at least 22-years-old
* A candidate for primary breast augmentation (general breast enlargement, post-lactational involution, asymmetry) or augmentation revision (previous augmentation with silicone-filled or saline-filled implants)
* Signs the Informed Consent
* Agrees to return device to Mentor if explant necessary
* Agrees to comply with follow-up procedures, including returning for all follow-up visits
* Patient is a US citizen with a Social Security Number

Exclusion Criteria:

* Subject is pregnant
* Has nursed a child within three months of study enrollment
* Been implanted with any silicone implant other than breast implants (e.g. silicone artificial joints or facial implants).
* Confirmed diagnosis of the following rheumatic diseases or syndromes: SLE, Sjogren's syndrome, scleroderma, polymyositis, or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyarthropathies, any other inflammatory arthritis, fibromyalgia, or chronic fatigue syndrome
* Currently has a condition that could compromise or complicate wound healing
* Has diagnosis of active cancer of any type
* Infection or abscess anywhere in the body
* Demonstrates tissue characteristics which are clinically incompatible with implant placement (e.g. tissue damage resulting from radiation, inadequate tissue, or compromised vascularity)
* Possesses any condition, or is under treatment for any condition which, in the opinion of the investigator and/or consulting physician(s), may constitute an unwarranted surgical risk
* Anatomic or physiologic abnormality which could lead to significant postoperative adverse events
* Demonstrates characteristics that are unrealistic/unreasonable with the risks involved with the surgical procedure
* Premalignant breast disease without a subcutaneous mastectomy
* Untreated or inappropriately treated breast malignancy, without mastectomy
* Are HIV positive
* Work for Mentor or the study doctor or are directly related to anyone that works for Mentor or the study doctor
* Implanted metal or metal devices, history of claustrophobia or other condition that would make a MRI scan prohibitive

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2024-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety will be determined by the incidence, severity, method of resolution, and duration for all adverse events on a per implant and per subject basis. | 10 years
Effectiveness will be determined by changes in chest circumference and bra and cup size. | 10 Years

SECONDARY OUTCOMES:
Effectiveness will also be determined by changes in validated Quality of Life instrument ratios. | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Kaveh Alizadeh, M.D., Principal Investigator — Garden City, NY; Joseph Bauer, M.D., Principal Investigator — Alpharetta, GA; Steven P. Bloch, M.D., Principal Investigator — Highland Park, IL; William R. Burden, M.D., Principal Investigator — Destin, FL; David Caplin, M.D., Principal Investigator — St. Louis, MO; Michael Cohen, M.D., Principal Investigator — Towson, MD; Steven Gitt, M.D., Principal Investigator — Phoenix, AZ; Mike E. Gonce, M.D., Principal Investigator — Oklahoma City, OK; Lawrence Gray, M.D., Principal Investigator — Portsmouth, NH; John Grossman, M.D., Principal Investigator — Denver, CO; W. Tracy Hankins, M.D., Principal Investigator — Lake Havasu City, AZ & Las Vegas, NV; Lars Enevoldsen, M.D., Principal Investigator — Modesto, CA; Neal Handel, M.D., Study Director — Medical Director - Sherman Oaks, CA; Jason Pozner, M.D., Principal Investigator — Boca Raton, FL; Cayce Rumsey, M.D., Principal Investigator — Ponte Vedra Beach, FL; Kimberly Short, M.D., Principal Investigator — Indianapolis, IN; Paul Silverstein, M.D., Principal Investigator — Oklahoma City, OK; Jon Trevisani, M.D., Principal Investigator — Maitland, FL; Douglas Wagner, M.D., Principal Investigator — Akron, OH; Simeon Wall Jr., M.D., Principal Investigator — Shreveport, LA; Wesley Wilson, M.D., Principal Investigator — Scottsdale, AZ; Richard Zienowicz, M.D., Principal Investigator — Providence, RI; Hilton Becker, MD, Principal Investigator — Boca Raton, FL; William Hedden, MD, Principal Investigator — Birmingham, AL; Jorge Perez, MD, Principal Investigator — Fort Lauderdale, FL; Marc Salzman, MD, Principal Investigator — Louisville, KY
Locations (1):
- Mentor Worldwide LLC, Santa Barbara, California, United States

REFERENCES:
- [Background] Bondurant, S., V.L. Ernster and R. Herdman, Eds. 2000. Safety of silicone breast implants. Committee on the Safety of Silicone Breast Implants, Division of Health Promotion and Disease Prevention, Institute of Medicine. Washington, D.C.: National Academy
- [Background] Holmich LR, Vejborg IM, Conrad C, Sletting S, Hoier-Madsen M, Fryzek JP, McLaughlin JK, Kjoller K, Wiik A, Friis S. Untreated silicone breast implant rupture. Plast Reconstr Surg. 2004 Jul;114(1):204-14; discussion 215-6. doi: 10.1097/01.prs.0000128821.87939.b5. PMID 15220594
- [Background] Holmich LR, Kjoller K, Vejborg I, Conrad C, Sletting S, McLaughlin JK, Fryzek J, Breiting V, Jorgensen A, Olsen JH. Prevalence of silicone breast implant rupture among Danish women. Plast Reconstr Surg. 2001 Sep 15;108(4):848-58; discussion 859-63. doi: 10.1097/00006534-200109150-00006. PMID 11547138
- [Background] Katzin WE, Centeno JA, Feng LJ, Kiley M, Mullick FG. Pathology of lymph nodes from patients with breast implants: a histologic and spectroscopic evaluation. Am J Surg Pathol. 2005 Apr;29(4):506-11. doi: 10.1097/01.pas.0000155145.60670.e4. PMID 15767806
- [Background] Berner I, Gaubitz M, Jackisch C, Pfleiderer B. Comparative examination of complaints of patients with breast-cancer with and without silicone implants. Eur J Obstet Gynecol Reprod Biol. 2002 Apr 10;102(1):61-6. doi: 10.1016/s0301-2115(01)00561-9. PMID 12039092
- [Background] Brown SL, Pennello G, Berg WA, Soo MS, Middleton MS. Silicone gel breast implant rupture, extracapsular silicone, and health status in a population of women. J Rheumatol. 2001 May;28(5):996-1003. PMID 11361228
- [Background] Holmich LR, Kjoller K, Fryzek JP, Hoier-Madsen M, Vejborg I, Conrad C, Sletting S, McLaughlin JK, Breiting V, Friis S. Self-reported diseases and symptoms by rupture status among unselected Danish women with cosmetic silicone breast implants. Plast Reconstr Surg. 2003 Feb;111(2):723-32; discussion 733-4. doi: 10.1097/01.PRS.0000041442.53735.F8. PMID 12560693
- [Background] Wolfe F, Anderson J. Silicone filled breast implants and the risk of fibromyalgia and rheumatoid arthritis. J Rheumatol. 1999 Sep;26(9):2025-8. PMID 10493686
- [Background] Brinton LA, Buckley LM, Dvorkina O, Lubin JH, Colton T, Murray MC, Hoover R. Risk of connective tissue disorders among breast implant patients. Am J Epidemiol. 2004 Oct 1;160(7):619-27. doi: 10.1093/aje/kwh272. PMID 15383405
- [Background] Janowsky EC, Kupper LL, Hulka BS. Meta-analyses of the relation between silicone breast implants and the risk of connective-tissue diseases. N Engl J Med. 2000 Mar 16;342(11):781-90. doi: 10.1056/NEJM200003163421105. PMID 10717013
- [Background] Lipworth L, Tarone RE, McLaughlin JK. Silicone breast implants and connective tissue disease: an updated review of the epidemiologic evidence. Ann Plast Surg. 2004 Jun;52(6):598-601. doi: 10.1097/01.sap.0000128087.51384.f9. PMID 15166995
- [Background] Tugwell P, Wells G, Peterson J, Welch V, Page J, Davison C, McGowan J, Ramroth D, Shea B. Do silicone breast implants cause rheumatologic disorders? A systematic review for a court-appointed national science panel. Arthritis Rheum. 2001 Nov;44(11):2477-84. doi: 10.1002/1529-0131(200111)44:113.0.co;2-q. PMID 11710703
- [Background] Williams HJ, Weisman MH, Berry CC. Breast implants in patients with differentiated and undifferentiated connective tissue disease. Arthritis Rheum. 1997 Mar;40(3):437-40. doi: 10.1002/art.1780400308. PMID 9082930
- [Background] Breiting VB, Holmich LR, Brandt B, Fryzek JP, Wolthers MS, Kjoller K, McLaughlin JK, Wiik A, Friis S. Long-term health status of Danish women with silicone breast implants. Plast Reconstr Surg. 2004 Jul;114(1):217-26; discussion 227-8. doi: 10.1097/01.prs.0000128823.77637.8a. PMID 15220596
- [Background] Fryzek JP, Signorello LB, Hakelius L, Feltelius N, Ringberg A, Blot WJ, McLaughlin JK, Nyren O. Self-reported symptoms among women after cosmetic breast implant and breast reduction surgery. Plast Reconstr Surg. 2001 Jan;107(1):206-13. doi: 10.1097/00006534-200101000-00034. PMID 11176625
- [Background] Kjoller K, Holmich LR, Fryzek JP, Jacobsen PH, Friis S, McLaughlin JK, Lipworth L, Henriksen TF, Hoier-Madsen M, Wiik A, Olsen JH. Self-reported musculoskeletal symptoms among Danish women with cosmetic breast implants. Ann Plast Surg. 2004 Jan;52(1):1-7. doi: 10.1097/01.sap.0000101930.75241.55. PMID 14676691
- [Background] Brinton LA, Lubin JH, Burich MC, Colton T, Brown SL, Hoover RN. Breast cancer following augmentation mammoplasty (United States). Cancer Causes Control. 2000 Oct;11(9):819-27. doi: 10.1023/a:1008941110816. PMID 11075871
- [Background] Bryant H, Brasher P. Breast implants and breast cancer--reanalysis of a linkage study. N Engl J Med. 1995 Jun 8;332(23):1535-9. doi: 10.1056/NEJM199506083322302. PMID 7739707
- [Background] Deapen DM, Bernstein L, Brody GS. Are breast implants anticarcinogenic? A 14-year follow-up of the Los Angeles Study. Plast Reconstr Surg. 1997 Apr;99(5):1346-53. doi: 10.1097/00006534-199704001-00022. PMID 9105362
- [Background] Herdman RC, Fahey TJ Jr. Silicone breast implants and cancer. Cancer Invest. 2001;19(8):821-32. doi: 10.1081/cnv-100107744. No abstract available. PMID 11768036
- [Background] Pukkala E, Boice JD Jr, Hovi SL, Hemminki E, Asko-Seljavaara S, Keskimaki I, McLaughlin JK, Pakkanen M, Teppo L. Incidence of breast and other cancers among Finnish women with cosmetic breast implants, 1970-1999. J Long Term Eff Med Implants. 2002;12(4):271-9. PMID 12627789
- [Background] Jakubietz MG, Janis JE, Jakubietz RG, Rohrich RJ. Breast Augmentation: Cancer Concerns and Mammography-A Literature Review. Plast Reconstr Surg. 2004 Jun;113(7):117e-22e. doi: 10.1097/01.PRS.0000122408.60459.92. PMID 27463401
- [Background] Miglioretti DL, Rutter CM, Geller BM, Cutter G, Barlow WE, Rosenberg R, Weaver DL, Taplin SH, Ballard-Barbash R, Carney PA, Yankaskas BC, Kerlikowske K. Effect of breast augmentation on the accuracy of mammography and cancer characteristics. JAMA. 2004 Jan 28;291(4):442-50. doi: 10.1001/jama.291.4.442. PMID 14747501
- [Background] McLaughlin JK, Lipworth L. Brain cancer and cosmetic breast implants: a review of the epidemiologic evidence. Ann Plast Surg. 2004 Feb;52(2):115-7. doi: 10.1097/01.sap.0000108560.71339.6c. PMID 14745257
- [Background] Cook LS, Daling JR, Voigt LF, deHart MP, Malone KE, Stanford JL, Weiss NS, Brinton LA, Gammon MD, Brogan D. Characteristics of women with and without breast augmentation. JAMA. 1997 May 28;277(20):1612-7. PMID 9168291
- [Background] Kjoller K, Holmich LR, Fryzek JP, Jacobsen PH, Friis S, McLaughlin JK, Lipworth L, Henriksen TF, Jorgensen S, Bittmann S, Olsen JH. Characteristics of women with cosmetic breast implants compared with women with other types of cosmetic surgery and population-based controls in Denmark. Ann Plast Surg. 2003 Jan;50(1):6-12. doi: 10.1097/00000637-200301000-00002. PMID 12545102
- [Background] Brinton LA, Lubin JH, Burich MC, Colton T, Brown SL, Hoover RN. Cancer risk at sites other than the breast following augmentation mammoplasty. Ann Epidemiol. 2001 May;11(4):248-56. doi: 10.1016/s1047-2797(00)00223-4. PMID 11306343
- [Background] Lugowski SJ, Smith DC, Bonek H, Lugowski J, Peters W, Semple J. Analysis of silicon in human tissues with special reference to silicone breast implants. J Trace Elem Med Biol. 2000 Apr;14(1):31-42. doi: 10.1016/S0946-672X(00)80021-8. PMID 10836532
- [Background] Kjoller K, Friis S, Signorello LB, McLaughlin JK, Blot WJ, Lipworth L, Mellemkjaer L, Winther JF, Olsen JH. Health outcomes in offspring of Danish mothers with cosmetic breast implants. Ann Plast Surg. 2002 Mar;48(3):238-45. doi: 10.1097/00000637-200203000-00002. PMID 11862026
- [Background] Signorello LB, Fryzek JP, Blot WJ, McLaughlin JK, Nyren O. Offspring health risk after cosmetic breast implantation in Sweden. Ann Plast Surg. 2001 Mar;46(3):279-86. doi: 10.1097/00000637-200103000-00014. PMID 11293521
- [Background] Hemminki E, Hovi SL, Sevon T, Asko-Seljavaara S. Births and perinatal health of infants among women who have had silicone breast implantation in Finland, 1967-2000. Acta Obstet Gynecol Scand. 2004 Dec;83(12):1135-40. doi: 10.1111/j.0001-6349.2004.00437.x. PMID 15548145
- [Background] Brinton LA, Lubin JH, Burich MC, Colton T, Hoover RN. Mortality among augmentation mammoplasty patients. Epidemiology. 2001 May;12(3):321-6. doi: 10.1097/00001648-200105000-00012. PMID 11337605
- [Background] Jacobsen PH, Holmich LR, McLaughlin JK, Johansen C, Olsen JH, Kjoller K, Friis S. Mortality and suicide among Danish women with cosmetic breast implants. Arch Intern Med. 2004 Dec 13-27;164(22):2450-5. doi: 10.1001/archinte.164.22.2450. PMID 15596635
- [Background] Koot VC, Peeters PH, Granath F, Grobbee DE, Nyren O. Total and cause specific mortality among Swedish women with cosmetic breast implants: prospective study. BMJ. 2003 Mar 8;326(7388):527-8. doi: 10.1136/bmj.326.7388.527. No abstract available. PMID 12623911
- [Background] Flassbeck D, Pfleiderer B, Klemens P, Heumann KG, Eltze E, Hirner AV. Determination of siloxanes, silicon, and platinum in tissues of women with silicone gel-filled implants. Anal Bioanal Chem. 2003 Feb;375(3):356-62. doi: 10.1007/s00216-002-1694-z. Epub 2003 Jan 28. PMID 12589499
- [Background] Stein, J., et al. 1999. In situ determination of the active catalyst in hydrosilylation reactions using highly reactive Pt(0) catalyst precursors. J. Am. Chem. Soc. 121(15):3693-3703
- [Background] Chandra, G., et al. 1987. A convenient and novel route to bis(alkyne)platinum(0) and other platinum(0) complexes from Speier's hydrosilylation catalyst. Organometallics. 6:191-2
- [Background] Lappert, M.F. and Scott, F.P.A. 1995. The reaction pathway from Speier's to Karstedt's hydrosilylation catalyst. J. Organomet. Chem. 492(2):C11-C13
- [Background] Lewis, L.N., et al. 1995. Mechanism of formation of platinum(0) complexes containing silicon-vinyl ligands. Organometallics. 14:2202-13